CLINICAL TRIAL: NCT00654511
Title: Dexmedetomidine for Immediate Perioperative Analgesia in Pediatric Patients Undergoing Tonsillectomy.
Acronym: DexT&A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Julia Finkel, MD, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3502; Agreement #10698
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Tonsillitis
Keywords: Dexmedetomidine,; fentanyl,; tonsillectomy; and adenoidectomy,
MeSH Terms: conditions — Tonsillitis | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fentanyl 1 (Active Comparator): Fentanyl 1 micrograms (mcg)/kilogram (kg)
  Interventions: Drug: Fentanyl
- Fentanyl 2 (Active Comparator): Fentanyl 2 micrograms (mcg)/kilogram (kg)
  Interventions: Drug: Fentanyl
- Dex 3 (Experimental): Dexmedetomidine 2 micrograms (mcg)/kilogram (kg)
  Interventions: Drug: Dexmedetomidine
- Dex 4 (Experimental): Dexmedetomidine 4 micrograms (mcg)/kilogram (kg)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 1mcg/kg, Intravenous (IV)
  Other Names: Actiq
  Arms: Fentanyl 1
Drug: Fentanyl — Fentanyl 2mcg/kg, Intravenous (IV)
  Other Names: Actiq
  Arms: Fentanyl 2
Drug: Dexmedetomidine — Dexmedetomidine, 2mcg/kg, Intravenous (IV)
  Other Names: Precedex
  Arms: Dex 3
Drug: Dexmedetomidine — Dexmedetomidine, 4mcg/kg Intravenous (IV)
  Other Names: Precedex
  Arms: Dex 4

SUMMARY:
The primary purpose of this study is:

1. To compare dexmedetomidine with fentanyl in terms of intra-operative hemodynamics and post-operative analgesia.
2. To determine an analgesic dose response relationship for dexmedetomidine.
3. Compare recovery characteristics of dexmedetomidine to fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* All of the following criteria must be met for the potential subject to be eligible for participation:

  1. The subject is 2 to 12 years of age
  2. The subject's American Society of Anesthesiologists physical status is ASA I or II (see appendix 1).
  3. The subject is scheduled for elective tonsillectomy with or without adenoidectomy surgery (procedures with myringotomy tube placement are allowed).
  4. The subject will be hospitalized overnight after surgery
  5. The subject's parent/legally authorized guardian has given written informed consent to participate; and where applicable, the subject has given appropriate assent to participate.

     Exclusion Criteria:
* The potential subject is NOT eligible for participation if any of the following exclusion criteria apply:

  1. The subject has a history or a family (parent or sibling) history of malignant hyperthermia
  2. The subject has known significant renal or hepatic disorders determined by medical history, physical examination or laboratory tests.
  3. The subject has a known or suspected allergy to opioid analgesics
  4. The subject is a pregnant or lactating female (if post-menarcheal, a negative pregnancy test must be confirmed prior to the planned surgery time (in AMSAC) consistent with current standard of care.
  5. The subject has history of. cardiovascular issues which would preclude the use of dexmedetomidine, (e.g. Down's Syndrome, dysrhthymias, conditions where hypotension is to be avoided).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Finkel, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Pestieau SR, Quezado ZM, Johnson YJ, Anderson JL, Cheng YI, McCarter RJ, Choi S, Finkel JC. High-dose dexmedetomidine increases the opioid-free interval and decreases opioid requirement after tonsillectomy in children. Can J Anaesth. 2011 Jun;58(6):540-50. doi: 10.1007/s12630-011-9493-7. Epub 2011 Apr 2. PMID 21461792

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl 1 Microgram/Kilogram Intravenous (IV): Fentanyl 1 microgram/kilogram IV given immediately after endotracheal intubation.
- Fentanyl 2 Micrograms/Kilogram Intravenous (IV): Fentanyl 2 micrograms/kilogram IV given immediately after endotracheal intubation
- Dexmedetomidine 2 Microgram/Kilogram Intravenous (IV): Dexmedetomidine 2mcg/kg given immediately after endotracheal intubation
- Dexmedetomidine 4 Micrograms/Kilogram Intravenous (IV): Dexmedetomidine 4mcg/kg given immediately after endotracheal intubation
Period: Overall Study
Arm/Group | Fentanyl 1 Microgram/Kilogram Intravenous (IV) | Fentanyl 2 Micrograms/Kilogram Intravenous (IV) | Dexmedetomidine 2 Microgram/Kilogram Intravenous (IV) | Dexmedetomidine 4 Micrograms/Kilogram Intravenous (IV)
Started | 26 | 25 | 25 | 25
Completed | 26 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl 1 Microgram/Kilogram Intravenous (IV) | Fentanyl 2 Micrograms/Kilogram Intravenous (IV) | Dexmedetomidine 2 Microgram/Kilogram Intravenous (IV) | Dexmedetomidine 4 Micrograms/Kilogram Intravenous (IV) | Total
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 25 | 25 | 25 | 101
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.17 (2.33) | 4.83 (2.45) | 5.17 (2.33) | 4.92 (2.27) | 4.77 (2.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 12 | 11 | 43
  Male | 17 | 14 | 13 | 14 | 58
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 25 | 25 | 101

OUTCOME MEASURES:

1. Primary Outcome: Time to First Morphine Dose
Description: Total minutes from study medication administration to time of first morphine dose.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fentanyl 1 Microgram/Kilogram IV | Fentanyl 2 Micrograms/Kilogram IV | Dexmedetomidine 2 Microgram/Kilogram IV | Dexmedetomidine 4 Micrograms/Kilogram IV
Number analyzed (Participants) | 26 | 25 | 25 | 25
minutes | 19 (24.8) | 43.7 (61.4) | 61.1 (89.5) | 137.6 (123.2)

2. Primary Outcome: Morphine Rescue
Description: Total morphine administered in the Post Anesthesia Care Unit (PACU)
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: micrograms/kilogram
Arm/Group | Fentanyl 1 Microgram/Kilogram Intravenous (IV) | Fentanyl 2 Micrograms/Kilogram Intravenous (IV) | Dexmedetomidine 2 Microgram/Kilogram Intravenous (IV) | Dexmedetomidine 4 Micrograms/Kilogram Intravenous (IV)
Number analyzed (Participants) | 26 | 25 | 25 | 25
micrograms/kilogram | 84 (37) | 95 (44) | 85 (37) | 59 (44)

ADVERSE EVENTS:
Arm/Group | Fentanyl 1 Microgram/Kilogram Intravenous (IV) | Fentanyl 2 Micrograms/Kilogram Intravenous (IV) | Dexmedetomidine 2 Microgram/Kilogram Intravenous (IV) | Dexmedetomidine 4 Micrograms/Kilogram Intravenous (IV)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes